CLINICAL TRIAL: NCT02812095
Title: Efficacy and Safety of Refeeding in Preterm Infants With Enterostomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Ee-Kyung Kim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: 1407-193-601
Record Dates: First submitted 2016-06-06; First posted 2016-06-24 (Estimated); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Enterostomy
MeSH Terms: interventions — RIFL protein, mouse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- The refeeding group (Experimental): Refeeding is initiated when 120mL/kg/day of enteral feed reaches or stoma loss exceeds more than 40ml/kg/day after operation.
  Interventions: Procedure: Refeeding
- The control group (No Intervention)

INTERVENTIONS:
Procedure: Refeeding — when amount of feeding reach to 120mL/kg a day,
  Other Names: extracorporeal stool transport
  Arms: The refeeding group

SUMMARY:
Refeeding is an extracorporeal stool transport from the proximal stoma end to the distal end of stoma. Refeeding may be beneficial in preventing malabsorption, electrolyte imbalance, cholestasis and atrophy of the distal intestine. Investigators are focused on evaluating the efficacy and safety of the practice of refeeding in preterm infants with enterostomy. Clinical data including weight gain, total parenteral nutrition (TPN) usage, and other laboratory findings will be collected. Serial citrulline levels during refeeding procedure and pathologic specimens of bowel (at the time of stoma closure) will be collected for evaluating bowel adaptation.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants who are less than 35 weeks gestational age at birth and get stomas after laparotomy

Exclusion Criteria:

* Congenital gastrointestinal malformation
* Blind pouch (after laparotomy)
* Refeeding procedure related infection
* Hemodynamic instability requiring inotropic or vasopressor agents (if the condition improves, the refeeding procedure can be restarted again)

Max Age: 35 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2014-08; Primary Completion 2019-12-11 (Actual); Study Completion 2020-04-16 (Actual)

PRIMARY OUTCOMES:
The change of citrulline level during the study period | up to 6 months of corrected age
  4 time points: at the time of full enteral feeding (>120 cc/kg/day), 4 weeks later after full enteral feeding, at the time of stoma closure operation, 12 weeks later after closure operation

SECONDARY OUTCOMES:
The pathologic findings after refeeding procedure | up to 8 weeks of corrected age
  villus height, crypt depth, mucosal thickening of pathologic specimens at the time of stoma closure operation
the number of days on parenteral nutrition | up to 8 weeks of corrected age
  the day of discontinuation of intravenous protein supplements
The weight gain | up to 6 months of corrected age
  differences in the admission weight Z-scores and end of study weight Z-scores
Adverse events during refeeding procedure | up to 8 weeks of corrected age
  bowel prolapse, enteral hemorrhage, abdominal distension, infection related stoma

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Lee ES, Kim EK, Shin SH, Jung YH, Song IG, Kim YJ, Kim HY, Choi YH, Moon KC, Kim B. Efficacy and safety of mucous fistula refeeding in preterm infants: an exploratory randomized controlled trial. BMC Pediatr. 2023 Mar 29;23(1):137. doi: 10.1186/s12887-023-03950-1. PMID 36991415